CLINICAL TRIAL: NCT06874153
Title: Non-Invasive Prediction of Necrotizing Enterocolitis in Preterm Neonates with Feeding Intolerance
Brief Title: Non-Invasive Prediction of Necrotizing Enterocolitis in Preterm Neonates with Feeding Intolerance Using Fecal Lipocalin-2 and Electrical Cardiometry
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Hassan, assistant lecturer, Ain Shams University
Other Study IDs: NEC prediction in preterm
Record Dates: First submitted 2025-03-02; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Feeding Intolerance in Preterm; NEC; Electrical Cardiometry; PreTerm Neonate
Keywords: preterm; NEC; Electrical Cardiometry; SMA flow; feeding intolerance in preterm; Fecal lipocalin-2
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- feeing intolerance group: Preterm neonates with gestational age ≤ 35 weeks, admitted to the NICU, started enteral feeding and were diagnosed as having feeding intolerance defined as stages IA and IB by modified bell's staging.
  Measuring superior mesenteric artery will be done on day 1 of diagnosis of feeding intolerance Cardiac output and delivery of oxygen to tissues (do2) will be measured on day 1 of the diagnosis of feeding intolerance, and follow-up will be done after 24 hours by electrical bioimpedance.
  Fecal Lipocalin-2 assessment in Stool sample

SUMMARY:
Prospective observational study to evaluate the efficiency of using electrical cardiometry in combination with fecal lipocalin-2 for prediction of NEC in preterm neonates with feeding intolerance

DETAILED DESCRIPTION:
Necrotizing enterocolitis is one of the most life-threatening conditions for premature infants in neonatal intensive care units (NICU) and is associated with severe intestinal inflammation and necrosis, which occurs in 5-16% of very low birth weight (VLBW) infants with a mortality rate of 20-50% and various long-term clinical sequelae for the survivors.

Although preterm intestinal epithelium is suggested to be predisposed to an exaggerated inflammatory response to the present microbiome, impaired mesenteric perfusion inducing bowel hypoxia and ischemia is suggested to be one of the factors playing a major role in the development of NEC.

Pathogenesis of NEC is multifactorial; however, one of the major factors is the disturbance in the end-organ blood ﬂow with early hypoperfusion and hypotension, predisposing for developing NEC in preterm neonates.

Electrical cardiometry (EC) is an impedance-based method that has been introduced for continuous noninvasive hemodynamic monitoring for cardiac output (CO) and DO2 in both term and preterm infants.

Clinical studies have shown that abnormal perfusion in the splanchnic circulation, particularly in the superior mesenteric artery (SMA), may have a role in the development of NEC in newborns so can be used for early diagnosis and evaluation of NEC progression.

Fecal lipocalin-2 (LCN2), also known as neutrophil gelatinase-associated lipocalin, is an anti-microbial molecule that was identified as a new robust biomarker for predicting NEC development in very low birth weight infants. LCN2 can predict half of the cases who will develop NEC in low birth weight preterms.

ELIGIBILITY:
Inclusion Criteria:

Preterm neonates with gestational age ≤ 35 weeks, admitted to NICU, started enteral feeding and diagnosed as having feeding intolerance defined as stage IA and IB by modified bell's staging

Exclusion Criteria:

1. Chromosomal anomaly or multiple congenital malformations.
2. Patient with surgical malformation of the intestinal tract (i.e. omphalocele, gastroschisis, malrotation, intestinal atresia)
3. Patient diagnosed as hypoxic ischemic encephalopathy.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates with gestational age ≤ 35 weeks, admitted to NICU, started enteral feeding and diagnosed as having feeding intolerance defined as stage IA and IB by modified bell's staging
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Electrical cardiometry for prediction of NEC in preterm neonates with feeding intolerance | 48 hours
  low cardiac output measured by electrical cardiometry predict NEC in preterm with feeding intolerance

SECONDARY OUTCOMES:
Fecal lipocalin-2 for prediction of NEC in preterm neonates with feeding intolerance | 48 hours
  High level of lipocalin-2 in stool sample predict NEC in preterm neonates with feeding intolerance
SMA flow in prediction of NEC in preterm neonates with feeding intolerance | 48 hours
  low flow through SMA predict NEC in preterm neonates with feeding intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain Shams university., Cairo, Abbasia, Egypt